CLINICAL TRIAL: NCT03738059
Title: Assessment of the Lowest Effective Dose of Dexmedetomidine in Attenuating the Hemodynamic Responses During Skull Pin Insertion in Patients Undergoing Elective Craniotomy: Randomized Control Study
Brief Title: The Lowest Effective Dose of Dexmedetomidine in Attenuating the Hemodynamic Responses During Skull Pin Insertion in Patients Undergoing Elective Craniotomy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mohammed AboelFadl, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17300238
Record Dates: First submitted 2018-11-05; First posted 2018-11-13 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Skull Pin Insertion
Keywords: Skull Pin Insertion; Dexmedetomidine; Hemodynamic Responses
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group I (placebo) (Placebo Comparator): will receive intravenous normal saline (NS)
  Interventions: Other: normal saline 0.9%
- group II (Dex 0.5) (Experimental): will receive intravenous Dex 0.5 mcg/kg
  Interventions: Drug: Dexmedetomidine Injection [Precedex]
- group III (Dex 0.25) (Experimental): will receive intravenous Dex 0.25 mcg/kg
  Interventions: Drug: Dexmedetomidine Injection [Precedex]
- group IV (Dex 0.2) (Experimental): will receive intravenous Dex 0.2 mcg/kg.
  Interventions: Drug: Dexmedetomidine Injection [Precedex]

INTERVENTIONS:
Drug: Dexmedetomidine Injection [Precedex] — will receive intravenous Dexmedetomidine
  Other Names: Dexmedetomidine
  Arms: group II (Dex 0.5); group III (Dex 0.25); group IV (Dex 0.2)
Other: normal saline 0.9% — will receive intravenous normal saline 0.9%
  Arms: group I (placebo)

SUMMARY:
Skull pins are used to immobilize the head during craniotomy. Fixation of skull pins causes acute hemodynamic changes which may affect cerebral autoregulation and hence cerebral blood flow. Therefore, maintenance of stable hemodynamic parameters during skull pin placement under general anesthesia is crucial to ensure adequate cerebral perfusion and prevention of acute rise of intracranial pressure

DETAILED DESCRIPTION:
Many different strategies have been used to minimize the hemodynamic responses to skull pin placement with varying results. Local anesthetic infiltration at pin application sites has been used but was always unsuccessful in obtunding the hemodynamic responses to skull pin placement. Dexmedetomidine, an alpha-2 adrenoceptor agonist, has been recently introduced as a sedative for patients on mechanical ventilation. In addition to its sedative effect; Dexmedetomidine has significant analgesic qualities and has been labeled as "analgesia-sparing". To the best of the investigator's knowledge, few studies investigated Dex use to suppress hemodynamic responses to skull pinning. The aim of the current study was to evaluate the lowest effective dose of Dexmedetomidine in attenuating the hemodynamic responses to skull pin placement for craniotomies. Lidocaine, administered subcutaneously at the head-holder pin sites, was more effective in preventing the blood pressure response to skull-pin than was deepening the level of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* 120 Adult patients,
* undergoing elective craniotomy
* ASA I and II patients

Exclusion Criteria:

* patients undergoing craniotomy for emergency surgery,
* raised ICP,
* obese patients (body mass index >30 kg/m2 for males and 28 kg/m2 for females),
* patients having systemic comorbidities (cardiac, renal, hepatic, and endocrinal),
* hypertensive patients (including those detected after admission),
* patients undergoing intracranial aneurysm clipping

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
arterial blood pressure change | before Skull Pin Insertion till 20 minutes
  systolic and diastolic blood pressure mmhg
heart rate change | before Skull Pin Insertion till 20 minutes
  heart rate beat/minute

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut governorate, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jamali S, Archer D, Ravussin P, Bonnafous M, David P, Ecoffey C. The effect of skull-pin insertion on cerebrospinal fluid pressure and cerebral perfusion pressure: influence of sufentanil and fentanyl. Anesth Analg. 1997 Jun;84(6):1292-6. doi: 10.1097/00000539-199706000-00022. PMID 9174309
- [Background] Levin R, Hesselvik JF, Kourtopoulos H, Vavruch L. Local anesthesia prevents hypertension following application of the Mayfield skull-pin head holder. Acta Anaesthesiol Scand. 1989 May;33(4):277-9. doi: 10.1111/j.1399-6576.1989.tb02907.x. PMID 2655365
- [Background] Geze S, Yilmaz AA, Tuzuner F. The effect of scalp block and local infiltration on the haemodynamic and stress response to skull-pin placement for craniotomy. Eur J Anaesthesiol. 2009 Apr;26(4):298-303. doi: 10.1097/EJA.0b013e32831aedb2. PMID 19262392
- [Background] Nagappa S, Kalappa S, Sridhara RB. Evaluation of the Hemodynamic Response of Intravenous Clonidine versus Ropivacaine Scalp Block to Insertion of Scalp Pins in Neurosurgical Patients. Anesth Essays Res. 2018 Jan-Mar;12(1):213-217. doi: 10.4103/0259-1162.194572. PMID 29628584
- [Background] Bharne S, Bidkar PU, Badhe AS, Parida S, Ramesh AS. Comparison of intravenous labetalol and bupivacaine scalp block on the hemodynamic and entropy changes following skull pin application: A randomized, open label clinical trial. Asian J Neurosurg. 2016 Jan-Mar;11(1):60-5. doi: 10.4103/1793-5482.165801. PMID 26889282